CLINICAL TRIAL: NCT00847353
Title: Normal Values of High Frequency ECG (HyperQ™) in Asymptomatic, Apparently Healthy Normal Weight vs. Obese Individuals and in Young and Masters Athletes
Brief Title: Normal Values of High Frequency ECG (HyperQ™) in Apparently Healthy Individuals and in Young and Masters Athletes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BSP Biological Signal Processing Ltd. (Industry)
Responsible Party: Prinicipal Investigator, The Ribstein Center for Sports Medicine and Research, Wingate
Other Study IDs: WIN_01
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Healthy; Asymptomatic; Obesity
Keywords: high frequency ECG; normal values; asymptomatic; obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of this study is to investigate depolarization characteristics represented by changes in HyperQ in asymptomatic, apparently healthy athletic and non-athletic individuals. We also aim to examine a subgroup of obese and non-obese subjects. The goal of the study is to establish normal HyperQ values in these populations and compare HyperQ values of age-matched athletic vs. non-athletic individuals of similar health status.

ELIGIBILITY:
Inclusion Criteria:

* An asymptomatic, apparently healthy patient performing a maximal exercise stress test

Exclusion Criteria:

* Contraindications for an exercise test
* Wolff-Parkinson-White (pre-excitation) syndrome
* Atrial Fibrillation or significant ventricular arrhythmia
* Treatment with Digoxin
* Pacemaker
* Pregnancy or suspected pregnancy
* QRS duration>120ms or other conduction delays

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample referred or self referred to stress testing
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-02 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Normal values for depolarization characteristics will be established for study groups | end of data collection

CONTACTS AND LOCATIONS:
Locations (1):
- The Ribstein Center for Sports Medicine and Research, Netanya, Israel